CLINICAL TRIAL: NCT00022451
Title: A Phase I Trial and Pharmacokinetic Study of R115777 in Pediatric Patients With Refractory Leukemia
Brief Title: Tipifarnib in Treating Young Patients With Refractory Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH); Children's Oncology Group (Network)
Masking: None | Purpose: Treatment
Other Study IDs: 010196; 01-C-0196C; COG-ADVL0116; NCI-1930; CDR0000068819; NCT00017888 (obsolete NCT alias)
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Leukemia
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; relapsing chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic myelogenous leukemia, BCR-ABL1 positive; childhood acute promyelocytic leukemia (M3); acute undifferentiated leukemia; juvenile myelomonocytic leukemia; childhood chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Biphenotypic, Acute; Leukemia, Myelomonocytic, Juvenile | interventions — tipifarnib

INTERVENTIONS:
Drug: tipifarnib

SUMMARY:
RATIONALE: Tipifarnib may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth.

PURPOSE: Phase I trial to study the effectiveness of tipifarnib in treating young patients who have refractory leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and toxicity profile of tipifarnib in pediatric patients with refractory leukemia.
* Determine the pharmacokinetics of this drug in these patients.
* Determine the toxicity profile of this drug in these patients.

Secondary

* Analyze the gene expression profile of leukemic blasts from these patients before and after treatment with this drug.
* Determine circulating levels of nerve growth factor and correlate these levels with clinical neurotoxicity from this drug in these patients.

OUTLINE: This is an open-label, dose-escalation study.

Patients receive oral tipifarnib every 12 hours on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of tipifarnib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity. At least 9 additional patients are treated at the MTD.

PROJECTED ACCRUAL: A total of 12-34 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed acute lymphoblastic leukemia, acute nonlymphoblastic leukemia, juvenile myelomonocytic leukemia (JMML), or chronic myelogenous leukemia (CML) in blast crisis

  * Refractory to standard curative therapy
  * Acute promyelocytic leukemia refractory to tretinoin and arsenic trioxide
  * Philadelphia chromosome-positive CML refractory to imatinib mesylate
* Greater than 25% blasts in bone marrow (M3 bone marrow) except for patients with JMML
* Active extramedullary disease allowed
* No active leptomeningeal leukemia

PATIENT CHARACTERISTICS:

Age:

* 21 and under

Performance status:

* Karnofsky 50-100% (over 10 years of age)
* Lansky 50-100% (10 years of age and under)

Life expectancy:

* Not specified

Hematopoietic:

* Not required to be normal

Hepatic:

* Bilirubin normal
* SGPT and SGOT normal
* No significant hepatic dysfunction
* No grade 3 or 4 liver function test results within the past month

Renal:

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min
* No significant renal dysfunction

Cardiovascular:

* No significant cardiac dysfunction

Pulmonary:

* No significant pulmonary dysfunction

Neurologic:

* No history of grand mal seizures grade 3 or greater except febrile seizures
* No persistent sensory or motor neuropathy greater than grade 2

Other:

* No clinically significant unrelated systemic illness
* No serious infection
* No organ dysfunction that would preclude study participation
* No requirement for total parenteral nutrition
* No known allergy to azoles (e.g., clotrimazole, fluconazole, ketoconazole, voriconazole)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 1 week since prior colony-stimulating factor therapy (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF]) except epoetin alfa
* At least 3 months since prior myeloablative therapy followed by bone marrow or stem cell transplantation
* No concurrent immunotherapy
* No concurrent GM-CSF or interleukin-11

Chemotherapy:

* At least 2 weeks since prior chemotherapy
* No concurrent intrathecal chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* At least 1 week since prior corticosteroids
* No concurrent corticosteroids (except for acute allergic reaction)

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* Recovered from nonhematologic toxicity of all prior therapy
* At least 1 week since prior retinoids
* No antacids (magnesium- or aluminum-containing formulations) within 2 hours of study drug
* No other concurrent investigational agents
* No concurrent retinoids
* No concurrent anticonvulsants

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2001-06; Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C. Widemann, MD, Study Chair — National Cancer Institute (NCI)
Locations (61):
- United States (56):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Shands Cancer Center at the University of Florida Health Science Center, Gainesville, Florida
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Scottish Rite Campus, Atlanta, Georgia
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Riley Children Cancer Center at Riley Hospital for Children, Indianapolis, Indiana
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Floating Hospital for Children, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey at Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Texas Children's Cancer Center, Houston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MBCCOP - South Texas Pediatrics, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (2):
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (3):
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec

REFERENCES:
- [Background] de Nigris F, Balestrieri ML, Napoli C. Targeting c-Myc, Ras and IGF cascade to treat cancer and vascular disorders. Cell Cycle. 2006 Aug;5(15):1621-8. doi: 10.4161/cc.5.15.3138. Epub 2006 Aug 1. PMID 16921263
- [Result] Widemann BC, Arceci RJ, Jayaprakash N, Fox E, Zannikos P, Goodspeed W, Goodwin A, Wright JJ, Blaney SM, Adamson PC, Balis FM. Phase 1 trial and pharmacokinetic study of the farnesyl transferase inhibitor tipifarnib in children and adolescents with refractory leukemias: a report from the Children's Oncology Group. Pediatr Blood Cancer. 2011 Feb;56(2):226-33. doi: 10.1002/pbc.22775. Epub 2010 Sep 21. PMID 20860038